CLINICAL TRIAL: NCT03204149
Title: Evaluation of Safety of Low Level Laser MC-8XL Device Treatment in Chronic Wounds
Brief Title: Evaluation of Safety of Low Level Laser Device Treatment in Chronic Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project termination
Sponsor: Medical Coherence LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BBL-0043-16
Record Dates: First submitted 2017-06-25; First posted 2017-06-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group will be treated with the MC-8XL laser device, emitting 808 nm laser beam with a green laser beam.
  Intervention: MC-8XL low level laser device and Standard wound care
  Interventions: Device: MC-8XL low level laser device and Standard wound care
- Control group (Sham Comparator): The control group will receive treatment with a sham laser device, emitting a low power green light with inactive Infrared (IR) laser for indication only.
  Intervention: Sham laser device and Standard wound care
  Interventions: Device: Sham laser device and Standard wound care

INTERVENTIONS:
Device: MC-8XL low level laser device and Standard wound care — The MC-8XL, a handheld Low Level Laser Therapy (LLLT) device, comprised of an infrared laser diode that generates wavelength of 808 nm and a green laser diode with a wavelength of 525 nm will be used to treat the experimental group.
  Along with the active LLLT, generally accepted standard wound care procedures will be used during the clinical trial by a qualified study nurse or doctor. These procedures will include wound cleaning and drying before irradiation with the laser device (sham or active). Each ulcer will be also assessed and debrided if needed.
  After irradiation, each ulcer will be dressed with saline gauze dressing and offloaded.
  Arms: Treatment group
Device: Sham laser device and Standard wound care — The Sham device is of similar appearance, emitting only green light for indication with a wavelength of 525 nm of a low power, with inactive IR laser which will be used in the Control group.
  Along with the sham device, the same generally accepted standard wound care procedures will be used.
  Arms: Control group

SUMMARY:
This is a randomized, double blind, placebo-controlled study to evaluate the safety of the low level laser MC-8XL device treatment in subjects with an unsuccessfully treated Diabetic Foot Ulcer (DFU) that has been present for at least 3 months.

Eligible subjects will be randomized to either Treatment group or Control group, following which, treatment of each subject will be provided by a qualified nurse at the clinic or in the home setting, everyday for up to 16 weeks.

Study assessments and adverse events monitoring will be also performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated Informed Consent Form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18 to 90
* Having a DFU of at least 3 months duration that had not improved after prior standard wound treatments
* HbA1c of <11.0
* Size of wounds: 1-10 cm2
* Having DFU of grades 2 or 3 according to Wagner's classification

Exclusion Criteria:

* Immeasurable wounds or wounds that are unsuited to this laser treatment (usually due to the wound's location, e.g. in the area between the toes).
* Uncontrolled Diabetes defined as an HbA1c of > 11.0
* Arterial insufficiency, Doppler vascular assessment (if needed- Ankle Brachial Index (ABI) < 0.6)
* Osteomyelitis in the bone.
* Photosensitivity
* Pregnancy
* Presence of any suspicious pre-cancerous or cancerous lesions, or having cancer.
* Being on medications that are immunosuppressive, may affect peripheral blood flow or may affect normal wound healing.
* Being on medications that might cause photosensitivity.
* Participation in any other clinical trial testing a device or drug.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Safety | On a weekly basis until the end of the 16 week treatment period
  assessing device related and general adverse events

SECONDARY OUTCOMES:
Wound Healing | On a weekly basis until the end of the 16 week treatment period or until complete wound closure
  Percent of wounds achieving complete wound closure, wound granulation and percent change in ulcer size/area

CONTACTS AND LOCATIONS:
Locations (1):
- Northern District Trauma & Wound Clinics Division, Maccabi Health Care Services, Haifa, Israel